CLINICAL TRIAL: NCT00131222
Title: Lungwena Child Nutrition Intervention Study-4, LCNI-4. A Single-centre Intervention Trial in Rural Malawi, Testing the Potency of RUTF Supplementation to Alleviate Moderate Malnutrition Among 6-17 Month Old Infants
Brief Title: Trial to Alleviate Malnutrition With Fortified Spread Given as a Food Supplement to Underweight Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tampere University (Other)
Collaborators: Academy of Finland (Other); Foundation for Paediatric Research, Finland (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SA-1200720-4
Record Dates: First submitted 2005-08-16; First posted 2005-08-17 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2007-04

CONDITIONS: Malnutrition
Keywords: Infant; Malnutrition; Sub-Saharan Africa; Treatment; Growth; Haemoglobin; Fortified spread; Food supplement
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Food supplement: fortified spread
Procedure: Food supplement: maize and soy flour

SUMMARY:
This study tests the hypothesis that underweight 6-17-month old infants receiving fortified spread as a food supplement for 12 weeks grow better during the supplementation than infants who are provided with maize-soy flour supplement.

DETAILED DESCRIPTION:
Childhood undernutrition is very common in rural Malawi, like in many other countries in Sub-Saharan Africa. Usually, undernutrition develops between 6 and 24 months of age. By two years of age, 30-50% of all children in rural Malawi are undernourished, predisposing them to subsequent morbidity, developmental delay and mortality. Urgent interventions are needed but the magnitude of the problem precludes a hospital-based management strategy. Therefore, emphasis must be on prevention and early home-based rehabilitation of children with mild-to-moderate malnutrition. However, the options for community based approaches are not as developed as those for institutional management of undernutrition.

The present study tests a recently developed nutrient -dense spread, ready-to use- therapeutic food (RUTF), which offers a potential solution to home based nutrition rehabilitation. The concept has previously been shown to work not only in therapeutic feeding of undernourished children in nutrition rehabilitation units in Malawi but also home based supplementation of undernourished children aged 42 to 60 months in Mangochi District, southern Malawi. In the present study the investigators will test the efficacy in growth promotion of this product when provided as a supplementary food to moderately underweight infants (defined as WAZ <-2) between 6 and 18 months of age.

The study will be conducted in Lungwena area, Mangochi District, rural Malawi. A total of 176 6-14 -month old infants will be enrolled and randomised to two groups receiving different daily food supplements for 12 weeks. Children in group one (control group) will receive 72g of fortified maize/soy flour and children in group 2 will receive 50g RUTF daily. The food supplements will be delivered to the participant's home at 3-weekly intervals.

All children will undergo medical and anthropometric examinations at 6-weekly intervals and disease symptoms monitoring every week. Dietary intake assessments will be conducted at 3 and 9 weeks after the onset of supplementation. A blood sample will be collected at the beginning and end of the study to measure blood haemoglobin and serum ferritin concentrations. At enrolment, children's HIV status will be screened with antibody-ELISA and confirmed with HIV PCR.

The impact of the dietary interventions will be primarily assessed by comparing weight gain in the two intervention groups. Secondary outcomes include length gain, increase in tibial length and changes in blood haemoglobin and serum ferritin concentration. The study will also produce descriptive data on morbidity and intake of foods during the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from at least one guardian
* Ages 6.00 months to 14.99 months
* Weight-for-age < -2 z-scores
* Availability during the period of the study
* Permanent resident of the area

Exclusion Criteria:

* WHZ < -3 z-scores or presence of oedema
* History of peanut allergy
* Severe illness warranting hospital referral
* Concurrent participation in another clinical trial with intervention to the child

Ages: 6 Months to 15 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 176
Dates: Start 2005-02; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Weight gain during the 12-week follow-up (in grams)

SECONDARY OUTCOMES:
Length gain during the study period (mm)
Tibial length gain during the study period (mm)
Change in blood haemoglobin concentration during the study period (g/l)
Change in serum ferritin concentration during the study period (µg/l)
Mean change in anthropometric indices (weight-for-age z-score [WAZ], weight-for-height z-score [WHZ] and height-for-age z-score [HAZ])

CONTACTS AND LOCATIONS:
Overall Officials: Per Ashorn, MD, PhD, Study Director — University of Tampere, Medical School; Kenneth M Maleta, MBBS, PhD, Principal Investigator — Kamuzu University of Health Sciences
Locations (1):
- College of Medicine, University of Malawi, Mangochi, Mangochi District, Malawi

REFERENCES:
- See also: College of Medicine home page — http://www.medcol.mw/